CLINICAL TRIAL: NCT00994682
Title: Long-term Role of Pioglitazone in Non-Alcoholic Fatty Liver Disease (NAFLD) in Type 2 Diabetes Mellitus (T2DM).
Brief Title: University of Texas H.S.C. San Antonio Pioglitazone in Non-Alcoholic Steatohepatitis Trial (UTHSCSA NASH Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The University of Texas at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20070654
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver Disease; Type 2 Diabetes Mellitus
Keywords: Additional relevant MeSH terms:; Hypoglycemic Agents; Physiological Effects of Drugs; Pharmacologic Actions; Pioglitazone
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pioglitazone (Active Comparator): After all patients receive dietary counseling at the research unit (CTSA), patients with prediabetes or type 2 diabetes mellitus (T2DM) and NASH will be started on pioglitazone (or placebo) in a randomized, double-blind,placebo-controlled study design. Pioglitazone will be given at 30 mg/day for the first 2 months and titrated to 45 mg/day thereafter (if well tolerated).
  Interventions: Drug: Pioglitazone study drug; Drug: Pioglitazone Open Label
- Placebo (Placebo Comparator): After dietary counseling to all patients at the research unit (CTSA), patients with prediabetes or type 2 diabetes mellitus (T2DM) and NASH will be started on pioglitazone (or placebo) in a randomized, double-blind,placebo-controlled study design. Pioglitazone will be given at 30 mg/day for the first 2 months and titrated to 45 mg/day thereafter (if well tolerated).
  Interventions: Drug: Placebo; Drug: Pioglitazone Open Label

INTERVENTIONS:
Drug: Pioglitazone study drug — 30 mg per day orally for 8 weeks, and if well tolerated, titrated to 45 mg per day until the end of 18 months
  Other Names: Actos (brand name), manufactured by Takeda Pharmaceuticals.
  Arms: Pioglitazone
Drug: Placebo — An oral tablet identical to pioglitazone will be given once daily but without active drug for 18 months.
  Arms: Placebo
Drug: Pioglitazone Open Label — Patients in both arms were placed open label pioglitazone for an additional 18 months after successfully completing the double-blind, placebo-controlled portion of the study design.
  Other Names: Actos (brand name), manufactured by Takeda Pharmaceuticals.

SUMMARY:
Obesity and Type 2 diabetes are creating a silent epidemic, Non-alcoholic fatty liver disease, which is a chronic liver disease associated with insulin resistance, impaired glucose intolerance, and hepatic fat accumulation. The thiazolidinedione pioglitazone improves glucose/lipid metabolism and histology in NASH by improving insulin resistance in the liver/peripheral/adipose tissues and reducing subclinical inflammation. The aim of this study is to assess the underlying mechanisms at the clinical and molecular level and the long-term efficacy and safety of pioglitazone in NASH in a multiethnic cohort of subjects (predominantly Hispanics, Caucasians and African-Americans - the most common ethnic groups locally) and examine the response including patients with normal glucose tolerance, impaired glucose tolerance or established type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
NASH is a disease characterized by elevated plasma aminotransferases and histopathological changes in liver characterized by hepatocellular steatosis, chronic inflammation and perisinusoidal fibrosis. NASH affects (~30-40%) of obese and type 2 diabetic subjects. While the pathogenesis of NASH is poorly understood, there is consensus that insulin resistance and its associated abnormalities in lipid metabolism play a key role in the development of liver fat accumulation. Insulin resistance in nonalcoholic steatohepatitis is frequently associated with chronic hyperinsulinemia, hyperglycemia, and an excessive supply of plasma free fatty acids to the liver. This in turn promotes hepatic lipogenesis. Pioglitazone, a thiazolidinedione (TZD), reverses these abnormalities by ameliorating insulin resistance in adipose tissue, liver and muscle. TZDs decrease excessive ectopic triglyceride accumulation in liver and muscle, reduce visceral fat, and redistribute fat to subcutaneous adipose stores. We have shown in a proof-of-concept 6-month study that pioglitazone is safe and effective for the treatment of T2DM. Patients with nonalcoholic steatohepatitis are also characterized by a low plasma adiponectin level. Thiazolidinediones increase plasma adiponectin levels, may activate AMP-activated protein kinase, stimulate hepatic/muscle fatty acid oxidation, and inhibit hepatic fatty acid synthesis in NASH nonalcoholic steatohepatitis. Thiazolidinediones also have antiinflammatory effects which are believed to be of value for therapy for NASH.

In order to evaluate this hypothesis, the investigators will treat for up to 36 months a group of patients with impaired (IGT) glucose tolerance and T2DM patients recruited from the University Hospital and medical school clinics and by newspaper add targeting the San Antonio and South Texas geographical area, with pioglitazone in a randomized, double-blinded, placebo-controlled trial. The primary endpoint will be liver histologic response assessed by liver biopsy performed at 18 and at 36 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to communicate meaningfully with the investigators and be legally competent to provide written informed consent.
2. Age range between 18 to 70 years (inclusive).
3. Female patients must be non-lactating and must either be at least one year post-menopausal, or be using adequate mechanical contraceptive precautions (i.e. intrauterine device, diaphragm with spermicide, condom with spermicide), or be surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy). Female patients who have undergone a hysterectomy are eligible for participation in the study. Female patients (except for those patients who have undergone a hysterectomy or a bilateral oophorectomy) are eligible only if they have a negative pregnancy test throughout the study period. Patients on oral contraceptives or an hormonal implant will be excluded (patches are acceptable as they deliver much lower estrogen systemically).
4. Participants must have the following laboratory values:

   * Hemoglobin ≥ 12 gm/dl in males, or ≥ 11 gm/dl in females,
   * WBC count ≥ 3,000/mm3
   * Neutrophil count ≥ 1,500/mm3
   * Platelets ≥ 100,000/mm3
   * Albumin ≥3.0 g/dl
   * Serum creatinine ≤ 1.8 mg/dl
   * Creatinine phosphokinase ≤ 2 times upper limit of normal
   * AST and ALT ≤ 3.0 times upper limit of normal
   * Alkaline phosphatase ≤ 2.5 times upper limit of normal
5. A diagnosis of NASH by liver biopsy performed within the past 6 months,

Exclusion Criteria:

1. Any cause of chronic liver disease other than NASH (such as -but not restricted to- alcohol or drug abuse, medication, chronic hepatitis B or C, autoimmune, hemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency).
2. Any clinical evidence or history of ascitis, bleeding varices, or spontaneous encephalopathy.
3. Current history of alcohol abuse (alcohol consumption greater than 20 grams of ethanol per day).
4. Prior surgical procedures to include gastroplasty, jejuno-ileal or jejunocolic bypass.
5. Prior exposure to organic solvents such as carbon tetrachloride.
6. Total parenteral nutrition (TPN) within the past 6 months.
7. Subjects with type 1 diabetes mellitus.
8. Patients on chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for 4 weeks before entry into the study. Patients on estrogens or other hormonal replacement therapy, tamoxifen, raloxifene, oral glucocorticoids or chloroquine will be excluded.
9. Patients with a history of clinically significant heart disease (New York Heart Classification greater than grade II), peripheral vascular disease (history of claudication), or diagnosed pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation).
10. Patients with severe osteoporosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cusi, M.D., Principal Investigator — University of Florida
Locations (1):
- Bartter Research Unit, Audie L Murphy VA Hospital, San Antonio, Texas, United States

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751
- [Derived] Bril F, Kalavalapalli S, Clark VC, Lomonaco R, Soldevila-Pico C, Liu IC, Orsak B, Tio F, Cusi K. Response to Pioglitazone in Patients With Nonalcoholic Steatohepatitis With vs Without Type 2 Diabetes. Clin Gastroenterol Hepatol. 2018 Apr;16(4):558-566.e2. doi: 10.1016/j.cgh.2017.12.001. Epub 2017 Dec 7. PMID 29223443
- [Derived] Cusi K, Orsak B, Bril F, Lomonaco R, Hecht J, Ortiz-Lopez C, Tio F, Hardies J, Darland C, Musi N, Webb A, Portillo-Sanchez P. Long-Term Pioglitazone Treatment for Patients With Nonalcoholic Steatohepatitis and Prediabetes or Type 2 Diabetes Mellitus: A Randomized Trial. Ann Intern Med. 2016 Sep 6;165(5):305-15. doi: 10.7326/M15-1774. Epub 2016 Jun 21. PMID 27322798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population of San Antonio, Texas, via newspaper advertisements and from the endocrinology and hepatology clinics at UTHSCSA and the Veterans Affairs Medical Center.
Pre-assignment Details: Once eligibility was met by histologically confirmed NASH, patients were randomized. The number of patients consented was 176, screen failed was 38, did not complete run-in phase was 37 (12 consent withdrawn, 9 lost to follow-up, 4 discontinued by PI decision, and 12 for other reasons). The remaining 101 patients were randomized.
Groups:
- Placebo: After all participants receive dietary counseling at the research unit (CTSA), patients with prediabetes or type 2 diabetes mellitus (T2DM) and NASH will be started on placebo (or pioglitazone) in a randomized, double-blind,placebo-controlled study design by the research pharmacy. Participants were prescribed a hypocaloric diet (500- kcal/d deficit from the calculated weight maintaining diet) and received placebo pills with identical physical characteristics and in identical bottles to pioglitazone pills.
- Pioglitazone: After dietary counseling to all patients at the research unit (CTSA), patients with prediabetes or T2DM and NASH will be started on pioglitazone (or placebo) in a randomized, double-blind,placebo-controlled study design. Participants were prescribed a hypocaloric diet (500- kcal/d deficit from the calculated weight maintaining diet) and received pioglitazone 30mg/d (titrated after 2 months to 45 mg/d).
Period: Double Bilnd
Arm/Group | Placebo | Pioglitazone
Started | 51 | 50
Completed | 42 | 41
Not Completed | 9 | 9
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 1 | 0
Period: Pioglitazone Open Label
Arm/Group | Placebo | Pioglitazone
Started | 42 | 41
Completed | 29 | 34
Not Completed | 13 | 7
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were prescribed a hypocaloric diet (500- kcal/d deficit from the calculated weight maintaining diet) and received placebo pills with identical physical characteristics and in identical bottles to pioglitazone pills. After 18 months of treatment, metabolic measurements (OGTT and euglycemic insulin clamp), DXA, 1H-MRS, and liver biopsy were repeated, at which point the medication code was disclosed to investigators and patients. Patients whose NASH resolved after 18 months were instructed to discontinue the study because pioglitazone treatment or a repeated liver biopsy were considered unethical and were not indicated, whereas those with persistent disease were invited to start open-label pioglitazone therapy, titrated as described for the other arm.
- Pioglitazone: Participants were prescribed a hypocaloric diet (500- kcal/d deficit from the calculated weight maintaining diet) and received pioglitazone 30mg/d (titrated after 2 months to 45 mg/d). After 18 months of treatment, metabolic measurements (OGTT and euglycemic insulin clamp), DXA, 1H-MRS, and liver biopsy were repeated, at which point the medication code was disclosed to investigators and patients. Patients initially assigned to pioglitazone were asked to continue at the same dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitazone | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11) | 52 (10) | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 35 | 36 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 31 | 68
  Not Hispanic or Latino | 14 | 19 | 33
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 99.2 (17.0) | 98.2 (16.5) | 98.7 (16.7)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (4.8) | 34.3 (4.8) | 34.4 (4.8)
Total body fat [Mean (Standard Deviation); unit: percentage of fat mass] — Measured by DXA
  percentage of fat mass | 34 (8) | 33 (7) | 33 (7)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dl] | 121 (27) | 124 (29) | 122 (28)
2-hour plasma glucose [Mean (Standard Deviation); unit: mg/dl] | 203 (64) | 211 (78) | 207 (71)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage] | 6.3 (1.0) | 6.4 (1.0) | 6.3 (1.0)
Fasting plasma insulin [Mean (Standard Deviation); unit: μU/mL] | 16 (12) | 15 (11) | 16 (11)
Fasting free fatty acids [Mean (Standard Deviation); unit: mmol/L] | 0.54 (0.19) | 0.49 (0.18) | 0.52 (0.19)
Use of diabetes medications [Number; unit: participants]
  Metformin | 17 | 19 | 36
  Sulfonylurea | 16 | 12 | 28
  Insulin | 6 | 5 | 11
Use of statins [Number; unit: participants] | 19 | 19 | 38
Plasma triglycerides [Mean (Standard Deviation); unit: mg/dl] | 179 (109) | 224 (171) | 201 (144)
Plasma total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 182 (42) | 187 (46) | 185 (44)
Plasma LDL-C [Mean (Standard Deviation); unit: mg/dl] | 109 (33) | 109 (44) | 109 (38)
Plasma HDL-C [Mean (Standard Deviation); unit: mg/dl] | 37 (9) | 36 (9) | 37 (9)
Plasma AST [Mean (Standard Deviation); unit: U/L] | 43 (22) | 47 (21) | 45 (22)
Plasma ALT [Mean (Standard Deviation); unit: U/L] | 57 (33) | 62 (33) | 60 (33)
NAFLD activity score (NAS) Liver histology [Mean (Standard Deviation); unit: score on a scale] — Steatosis: 0 = <5%; 1 = 5-33%; 2 = >33-66%; 3 = >66%. Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x.
  Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning.
  Total NAS score represents the sum of scores for steatosis, lobular inflammation, and ballooning. It is assessed on a scale of 0-8, with higher scores indicating more severe disease.
  score on a scale | 4.5 (1.2) | 4.5 (1.5) | 4.5 (1.3)
Steatosis grade [Mean (Standard Deviation); unit: units on a scale] — Steatosis: grade 0 = <5% of liver fat by histology; grade 1 = 5-33% liver fat; grade 2 = >33-66% liver fat; 3 = >66% liver fat, with higher scores indicating more severe disease.
  units on a scale | 1.9 (0.8) | 2.0 (0.8) | 2.0 (0.8)
Inflammation grade [Mean (Standard Deviation); unit: units on a scale] — Lobular Inflammation: grade 0 = No foci of inflammatory cells in the liver histology; grade 1 = <2 foci/200x; grade 2 = 2-4 foci/200x, grade 3 = >4 foci/200x, with higher scores indicating more severe disease.
  units on a scale | 1.7 (0.5) | 1.7 (0.6) | 1.7 (0.5)
Ballooning grade [Mean (Standard Deviation); unit: units on a scale] — Hepatocyte Ballooning: 0 = No ballooning cells observed in liver histology; 1 = Few balloon cells; 2 = Many cells/prominent ballooning, with higher scores indicating more severe disease.
  units on a scale | 0.9 (0.4) | 0.8 (0.4) | 0.9 (0.4)
Fibrosis stage [Mean (Standard Deviation); unit: units on a scale] — Fibrosis: 0 = No fibrosis in liver histology; 1 = Perisinusoidal or periportal, 1A = Mild, zone 3, perisinusoidal "delicate" fibrosis; 1B = Moderate, zone 3, perisinusoidal "dense" fibrosis; 1C = Portal/periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis, with higher scores indicating more severe disease.
  units on a scale | 0.9 (0.9) | 1.1 (1.1) | 1.0 (1.0)
Diagnosis of definite NASH [Number; unit: participants] | 45 | 42 | 87

OUTCOME MEASURES:

1. Primary Outcome: Liver Histology (Using Kleiner et al Criteria, Hepatology 2005)
Description: Number of patients with reduction of at least 2 points in the nonalcoholic fatty liver disease activity score (NAS) (with reduction in at least 2 different histological categories) without worsening of fibrosis. NAS is the sum of the separate scores for steatosis (0-3), hepatocellular ballooning (0-2) and lobular inflammation (0-3), and ranges from 0-8 .
  The scoring system is based on the following grading:
  Steatosis: 0 = <5%; 1 = 5-33%; 2 = >33-66%; 3 = >66%. Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x. Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning. Fibrosis: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis.
Time Frame: At 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
Participants | 9 | 29

2. Secondary Outcome: Number of Participants With Resolution of NASH
Description: Resolution of NASH was defined as absence of NASH after 18 months of therapy in patients with definite NASH (presence of zone 3 accentuation of macrovesicular steatosis of any grade, hepatocellular ballooning of any degree, and lobular inflammatory infiltrates of any amount) at baseline.
Time Frame: Month 18
Population: Multiple imputation was used to impute missing histologic data for patients who did not complete 18 months of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
Participants | 10 | 26

3. Secondary Outcome: Mean Individual Histological Scores
Description: Mean change in individual scores compared to baseline. Steatosis: 0 = <5%; 1 = 5-33%; 2 = >33-66%; 3 = >66%. Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x. Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning. Fibrosis: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis
Time Frame: Baseline and Month 18
Population: Multiple imputation was used to impute missing histologic data for patients who did not complete 18 months of therapy.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
units on a scale
  Steatosis | -0.2 [-1.8 to 1.4] | -1.1 [-2.7 to 0.5]
  Inflammation | -0.1 [-1.7 to 1.5] | -0.6 [-2.2 to 1.0]
  Ballooning | -0.2 [-1.8 to 1.4] | -0.6 [-2.2 to 1.0]
  Fibrosis | 0 [-1.568 to 1.568] | -0.5 [-2.1 to 1.1]

4. Secondary Outcome: Individual Histological Scores
Description: Number of patients with improvement of at least 1 grade in each of the histological parameters.
  Steatosis: 0 = <5%; 1 = 5-33%; 2 = >33-66%; 3 = >66%. Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x. Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning. Fibrosis: 0 = None; 1 = Perisinusoidal or periportal, 1A = Mild, zone 3, perisinusoidal "delicate" fibrosis; 1B = Moderate, zone 3, perisinusoidal "dense" fibrosis; 1C = Portal/periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis
Time Frame: Month 18
Population: Multiple imputation was used to impute missing histologic data for patients who did not complete 18 months of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
Participants
  Steatosis | 13 | 35
  Inflammation | 11 | 25
  Ballooning | 12 | 25
  Fibrosis | 13 | 20

5. Secondary Outcome: Mean Individual Histological Scores
Description: Steatosis: 0 = <5%; 1 = 5-33%; 2 = >33-66%; 3 = >66%. Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x. Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning. Fibrosis: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis
Time Frame: Month 36
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 29 | 34
units on a scale
  Steatosis | 1.56 [1.22 to 1.89] | 0.97 [0.67 to 1.27]
  Inflammation | 1.30 [0.80 to 1.51] | 0.81 [0.60 to 1.03]
  Ballooning | 0.33 [0.14 to 0.52] | 0.22 [0.07 to 0.37]
  Fibrosis | 0.89 [0.49 to 1.29] | 0.66 [0.32 to 0.99]

6. Secondary Outcome: Liver Transaminases (AST and ALT).
Time Frame: 18 and 36 months
Population: Data include 101 observations at baseline (51 in the placebo group and 50 in the pioglitazone group), 83 at month 18 (42 and 41, respectively), and 63 at month 36 (29 and 34, respectively).
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
U/L
  ALT at month 18 | 44 (33) | 27 (12)
  AST at month 18 | 38 (31) | 29 (10)
  ALT at month 36 | 32 (17) | 27 (13)
  AST at month 36 | 30 (10) | 27 (8)

7. Secondary Outcome: Liver Fat by Magnetic Resonance and Spectroscopy (MRS).
Description: Liver fat content was calculated as the fat fraction: 100*(area under the curve [AUC] of fat peak / [AUC of fat peak + AUC of water peak]).
Time Frame: 18 months
Population: Data include 101 observations at baseline (51 in the placebo group and 50 in the pioglitazone group) and 83 at month 18 (42 and 41, respectively).
Measure: Mean (Standard Deviation); unit: percentage of fat in liver
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 42 | 41
percentage of fat in liver | 11 (7) | 7 (5)

8. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Homeostatic model assessment of insulin resistance (HOMA-IR) is a method for assessing insulin resistance (IR) from basal fasting plasma glucose (FPG) and fasting plasma insulin (FPI). It is calculated as (FPG x FPI)/405.
Time Frame: 18 and 36 months
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Arbitrary units
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
Arbitrary units
  HOMA-IR month 18: number analyzed (Participants) | 42 | 41
  HOMA-IR month 18 | 4.3 [2.9 to 5.7] | 1.4 [1.0 to 1.8]
  HOMA-IR month 36: number analyzed (Participants) | 29 | 34
  HOMA-IR month 36 | 2.3 [1.4 to 3.3] | 1.6 [1.1 to 2.1]

9. Secondary Outcome: Hepatic Insulin Sensitivity
Description: Suppression of endogenous glucose production (Supp EGP) by low dose insulin (i.e., percentage of reduction of EGP with low dose insulin infusion compared to the baseline state). This was calculated as: 100*((EGP without insulin - EGP with insulin infusion)/EGP without insulin). All measurements are obtained at the same time point during an euglycemic insulin clamp.
Time Frame: 18 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: % of suppression of EGP
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 42 | 41
% of suppression of EGP | 37.7 [30.6 to 44.7] | 55.3 [47.2 to 63.5]

10. Secondary Outcome: Adipose Tissue Insulin Sensitivity
Description: Suppression of free fatty acids by low dose insulin (i.e., percentage of reduction of plasma FFA with low dose insulin infusion compared to the baseline state). This was calculated as: 100*((plasma FFA without insulin - plasma FFA with insulin infusion)/plasma FFA without insulin). All measurements are obtained at the same time point during an euglycemic insulin clamp.
Time Frame: 18 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: % of suppression of FFA
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 42 | 41
% of suppression of FFA | 46.1 [38.8 to 53.5] | 65.9 [60.6 to 71.3]

11. Secondary Outcome: Skeletal Muscle Insulin Sensitivity
Description: Rate of glucose disappearance (Rd) during high-dose insulin infusion. The rate of plasma glucose disappearance was calculated using Steele's non-steady-state equation.
Time Frame: 18 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: mg/kgLBM/min
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 42 | 41
mg/kgLBM/min | 5.4 [4.6 to 6.2] | 9.6 [8.2 to 11.1]

12. Secondary Outcome: Body Mass Index (BMI)
Time Frame: Months 18 and 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
kg/m^2
  BMI Month 18: number analyzed (Participants) | 42 | 41
  BMI Month 18 | 34.6 (5.0) | 34.6 (4.8)
  BMI Month 36: number analyzed (Participants) | 29 | 34
  BMI Month 36 | 36.7 (5.7) | 35.2 (4.8)

13. Secondary Outcome: Total Body Fat
Description: Total body fat measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: Months 18
Population: Data include 101 observations at baseline (51 in the placebo group and 50 in the pioglitazone group), 83 at month 18 (42 and 41, respectively).
Measure: Mean (Standard Deviation); unit: Percentage of body weight that is fat
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 42 | 41
Percentage of body weight that is fat | 36 (8) | 36 (7)

14. Secondary Outcome: Plasma Biomarkers Relevant to Hepatic Inflammation, Apoptosis and Fibrosis (Adiponectin).
Time Frame: 18 and 36 months
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
μg/ml
  Adiponectin month 18: number analyzed (Participants) | 42 | 41
  Adiponectin month 18 | 9.1 [7.1 to 11.1] | 22.8 [19.0 to 26.5]
  Adiponectin month 36: number analyzed (Participants) | 29 | 34
  Adiponectin month 36 | 24.0 [14.5 to 33.5] | 24.2 [18.6 to 29.8]

15. Secondary Outcome: Plasma Biomarkers Relevant to Hepatic Inflammation, Apoptosis and Fibrosis (CK-18).
Time Frame: 18 and 36 months
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Placebo | Pioglitazone
Number analyzed (Participants) | 51 | 50
U/L
  CK-18 month 18: number analyzed (Participants) | 42 | 41
  CK-18 month 18 | 314 [247 to 381] | 186 [133 to 238]
  CK-18 month 36: number analyzed (Participants) | 29 | 34
  CK-18 month 36 | 245 [184 to 305] | 151 [114 to 189]

16. Secondary Outcome: Prevention of the Onset of T2DM and/or Reversal From IFG/IGT to NGT in Non-diabetics.
Description: Number of patients developing T2DM and number of patients regressing to NGT among patients with prediabetes (IFG/IGT).
Time Frame: 18 months
Population: Only patients with prediabetes are included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 26 | 23
Participants
  Patients developing T2DM | 1 | 2
  Patients regressing to NGT | 10 | 1

17. Secondary Outcome: Osteoporotic Fractures
Description: Number of patients with osteoporotic fractures
Time Frame: 18 and 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 50 | 51
Participants | 0 | 0

18. Secondary Outcome: Molecular Pathways of Liver Glucose and Lipid Signaling; Inflammatory Pathways; Oxidative Stress; Other.
Time Frame: At 18 (2nd liver biopsy) and 36 (3rd liver biopsy) months.
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Bone Mineral Density
Description: Bone mineral density measured at the levels of spine, femoral neck, hip, and wrist by DXA.
Time Frame: 18 and 36 months
Population: Data analysis included 78 patients at month 18 and 62 at month 36 (based on DXA availability).
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 39 | 39
g/cm^2
  Spine BMD at month 18 | 1.04 (0.17) | 1.10 (0.17)
  Femoral Neck BMD at month 18 | 0.84 (0.13) | 0.86 (0.12)
  Hip BMD at month 18 | 1.05 (0.13) | 1.05 (0.13)
  Wrist BMD at month 18 | 0.76 (0.08) | 0.78 (0.09)
  Spine BMD at month 36: number analyzed (Participants) | 34 | 28
  Spine BMD at month 36 | 1.06 (0.14) | 1.10 (0.21)
  Femoral Neck BMD at month 36: number analyzed (Participants) | 34 | 28
  Femoral Neck BMD at month 36 | 0.84 (0.14) | 0.84 (0.12)
  Hip BMD at month 36: number analyzed (Participants) | 34 | 28
  Hip BMD at month 36 | 1.02 (0.12) | 1.06 (0.16)
  Wrist BMD at month 36: number analyzed (Participants) | 34 | 28
  Wrist BMD at month 36 | 0.75 (0.08) | 0.77 (0.09)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire study (36 months for each patient).
Groups:
- Placebo (First 18 Months): Participants were prescribed a hypocaloric diet (500- kcal/d deficit from the calculated weight maintaining diet) and received placebo pills with identical physical characteristics and in identical bottles to pioglitazone pills.
- Pioglitazone (First 18 Months): Participants were prescribed a hypocaloric diet (500- kcal/d deficit from the calculated weight maintaining diet) and received pioglitazone 30mg/d (titrated after 2 months to 45 mg/d).
- Placebo (PIO Open-label): After being randomized to placebo for the first 18 months, patients whose NASH resolved after 18 months were instructed to discontinue the study because pioglitazone treatment or a repeated liver biopsy were considered unethical and were not indicated, whereas those with persistent disease were invited to start open-label pioglitazone therapy, titrated as described for the other arm.
- Pioglitazone (Months 18-36): After 18 months of treatment, metabolic measurements (OGTT and euglycemic insulin clamp), DXA, 1H-MRS, and liver biopsy were repeated, at which point the medication code was disclosed to investigators and patients. Patients initially assigned to pioglitazone were asked to continue at the same dose.
Arm/Group | Placebo (First 18 Months) | Pioglitazone (First 18 Months) | Placebo (PIO Open-label) | Pioglitazone (Months 18-36)
Serious Adverse Events (participants affected / at risk) | 5/51 | 5/50 | 10/36 | 9/40
Other Adverse Events (participants affected / at risk) | 7/51 | 15/50 | 12/36 | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (First 18 Months) (N=51) | Pioglitazone (First 18 Months) (N=50) | Placebo (PIO Open-label) (N=36) | Pioglitazone (Months 18-36) (N=40)
Atypical chest pain (Cardiac disorders) | 1 | 1 | 0 | 2
Pulmonary thromboembolism (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colelithiasis (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diagnosis of adrenal carcinoma (Endocrine disorders) | 0 | 0 | 1 | 0
Dissociative amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Ovarian cyst rupture (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Diagnosis of prostate cancer (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urine retention (Renal and urinary disorders) | 0 | 0 | 2 | 0
Kidney stones (Renal and urinary disorders) | 0 | 0 | 0 | 2
Biopsy-related (Surgical and medical procedures) | 3 | 1 | 1 | 1
Motor vehicle accident (Social circumstances) | 0 | 1 | 0 | 0
Concussion (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (First 18 Months) (N=51) | Pioglitazone (First 18 Months) (N=50) | Placebo (PIO Open-label) (N=36) | Pioglitazone (Months 18-36) (N=40)
Chronic lower limb edema (Vascular disorders) | 3 | 11 | 5 | 0
Hypoglycemia (Endocrine disorders) | 4 | 4 | 7 | 10

LIMITATIONS AND CAVEATS:
The single-center nature of this study is a limitation that calls for additional work from a larger, longer-term (>3 years), multicenter trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No